CLINICAL TRIAL: NCT04282213
Title: Comparison of the TOFCuff Monitor Versus Electromyography in Neuromuscular Monitoring
Brief Title: Neuromuscular Monitoring:TOFCuff Versus EMG
Status: Completed | Type: Observational
Sponsor: Servei Central d'Anestesiologia (Other)
Responsible Party: Principal Investigator, Lorena Silva Gil, Principal Investigator, Servei Central d'Anestesiologia
Other Study IDs: NMT2020
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control samples: For each case, neuromuscular measurements gathered with GE CARESCAPE B450 monitor (E-NMT module).
- Case samples: For each case, neuromuscular measurements gathered with TOFCuff monitor.

SUMMARY:
Mechanomyography (MMG) is considered the gold-standard for neuromuscular blockade (NMB) monitoring. However, it is quite bulky and difficult to use on a routine basis. Therefore, alternative methods like Acceleromyography (AMG), Electromyography (EMG) and the TOF-CUFF method have been developed. The aim of this study was to compare the TOF-Cuff monitor and Electromyography (EMG-NMT module with the CARESCAPE B450 monitor) data following rocuronium-induced neuromuscular blockade and its reversal.

DETAILED DESCRIPTION:
Neuromuscular relaxation of the patient during surgery is necessary for multiple reasons, such as facilitating intubation or improving the effectiveness of some surgical procedures. Premature extubation of the patient without having achieved a complete recovery of the NMB can have deleterious consequences, increasing postoperative complications, especially those related to the respiratory system. Given this, current guidelines of good clinical practice recommend the monitoring of pharmacologically induced NMB during general anesthesia. In addition, monitoring allows confirmation of optimum relaxation before intubation, and allows for control over re-dose administration and recovery of NMB upon awakening from general anesthesia.

There are different methods of quantitative monitoring of NMB. The TOF-CUFF monitor uses a method based on a traditional pressure cuff that incorporates stimulation electrodes. The placement of the cuff which aligns the stimulation electrodes on the path of the brachial plexus at the humeral level allows to evaluate the muscular response evoked from the changes in the cuff pressure, generated by the muscular contraction after the electrical stimulus. Its main advantage is that monitoring of the NMB is included within the pressure cuff itself, which is always used in any anesthetic act. Then, when the pressure cuff is placed, monitoring of the NMB is easily established. This specific design facilitates the task of anesthesiologists because they do not have to perform any additional preparation for the monitoring of NMB.

The TOF-CUFF monitor has been validated regarding the mechanomyography, which is considered the gold-standard for the monitoring of NMB. The main objective of the study is to compare the values of NMB measured with the TOF-CUFF monitor with NMB values measured with the CARESCAPE B450 monitor during the pharmacologically induced NMB and evaluate the degree of equivalence in different situations. Secondary objective is to verify that the design for joint monitoring of the NMB and NIBP in the TOF-CUFF monitor does not affect the independent measure of the two variables.

Prospective, single-center, open and controlled observational clinical study. The study is aimed to be conducted with 40 patients aged between 18 and 65 years.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Patients who give their written informed consent
* Elective surgery under general anesthesia that according to the anesthetic plan muscle relaxants will be administered

Exclusion Criteria:

* Patients who refuse to give their informed consent
* Patients who present any of the contraindications for the devices used in the study
* Patients who are participating or have participated in a clinical trial during the 4 weeks prior to inclusion
* Women of childbearing age who do not use effective contraceptive methods, pregnant women, with suspicion of pregnancy or breast-feeding
* Patients with the following criteria: upper limb peripheral vascular pathologies, a difficult airway, myasthenia gravis and other neuromuscular diseases, use of medication that may alter NMT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients American Society of Anesthesiologist (ASA) I-II, between 18-65 years and scheduled for elective surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
TOFR (Train Of Four Ratio) | Baseline
  For this measurement, patient is stimulated with four twitches at a known stimulation current. Each twitch is performed every 500ms. The neuromuscular response for each twitch is gathered. Train Of Four ratio consists of the weighting of the fourth stimulus against the first stimulus.
  It can be calculated also as a percentage.
Counts | Baseline
  When performing the Train Of Four (TOF) measurement, count of the twitches that are higher than 0.
PTC | Baseline
  Once patient is in a deep neuromuscular blockade, all twitches from Train Of Four (TOF) measurement are 0. In order to evaluate the neuromuscular response, Post Tetanic Count (PTC) measurement is performed.
  PTC is splitted in two steps. First, during 5 seconds a tetanic stimulation is performed at 50Hz. If no response is elicited, after a pause of 3 seconds 15 single-twitch stimualtion at 1Hz are performed. PTC value is the count of the single-twitches that are higher than 0.
T1 | Baseline
  For Train Of Four (TOF) measurement, amplitude of the first neuromuscular stimulation response. Units depend on the measurement techniques.
T2 | Baseline
  For Train Of Four (TOF) measurement, amplitude of the second neuromuscular stimulation response. Units depend on the measurement techniques.
T3 | Baseline
  For Train Of Four (TOF) measurement, amplitude of the third neuromuscular stimulation response. Units depend on the measurement techniques.
T4 | Baseline
  For Train Of Four (TOF) measurement, amplitude of the fourth neuromuscular stimulation response. Units depend on the measurement techniques.
PID | Baseline
  Diastolic pressure in mmHg
PIS | Baseline
  Systolic pressure in mmHg
PIM | Baseline
  Mean pressure in mmHg

SECONDARY OUTCOMES:
Temperature | Baseline
  Patient temperature on the palm hand

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Silva Gil, MD, Principal Investigator — Servei d'Anestesiologia Centro Médico Teknon
Locations (1):
- Centro Médico Teknon, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naguib M, Kopman AF, Lien CA, Hunter JM, Lopez A, Brull SJ. A survey of current management of neuromuscular block in the United States and Europe. Anesth Analg. 2010 Jul;111(1):110-9. doi: 10.1213/ANE.0b013e3181c07428. Epub 2009 Nov 12. PMID 19910616
- [Background] Veiga Ruiz G, Garcia Cayuela J, Orozco Montes J, Parreno Caparros M, Garcia Rojo B, Aguayo Albasini JL. Monitoring intraoperative neuromuscular blockade and blood pressure with one device (TOF-Cuff): A comparative study with mechanomyography and invasive blood pressure. Rev Esp Anestesiol Reanim. 2017 Dec;64(10):560-567. doi: 10.1016/j.redar.2017.03.013. Epub 2017 Jun 27. English, Spanish. PMID 28662770
- [Background] Rodiera J, Serradell A, Alvarez-Gomez JA, Aliaga L. The cuff method: a pilot study of a new method of monitoring neuromuscular function. Acta Anaesthesiol Scand. 2005 Nov;49(10):1552-8. doi: 10.1111/j.1399-6576.2005.00777.x. PMID 16223405
- [Background] Checketts MR, Jenkins B, Pandit JJ. Implications of the 2015 AAGBI recommendations for standards of monitoring during anaesthesia and recovery. Anaesthesia. 2017 Jan;72 Suppl 1:3-6. doi: 10.1111/anae.13736. No abstract available. PMID 28044335
- [Background] Dahaba AA, von Klobucar F, Rehak PH, List WF. The neuromuscular transmission module versus the relaxometer mechanomyograph for neuromuscular block monitoring. Anesth Analg. 2002 Mar;94(3):591-6; table of contents. doi: 10.1097/00000539-200203000-00021. PMID 11867381